CLINICAL TRIAL: NCT04901026
Title: Satisfaction With an In-house Developed Nasal Foreign Body Removal Manikin: A Randomized-controlled Trial
Brief Title: Satisfaction With an In-house Developed Nasal Foreign Body Removal Manikin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Pittayapon Pitathawatchai, Assistant professor, Prince of Songkla University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 64-019-13-1
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Satisfaction; Consumer Satisfaction
Keywords: manikin; nasal foreign body
MeSH Terms: conditions — Personal Satisfaction; Consumer Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An in-house manikin (Active Comparator): Participants use an in-house manikin
  Interventions: Other: An in-house manikin
- A manikin in market (Sham Comparator): Participants use a manikin from market
  Interventions: Other: An in-house manikin

INTERVENTIONS:
Other: An in-house manikin — Participants obtain an in-house manikin

SUMMARY:
To overcome the issues regarding training in real persons, using a simulated manikin instead of an actual patient or simulated patient is another option with consideration to the training able to be held at any time periods and no issues about minor or serious complications needed to be concerned with. The aim of this study is to devise a low-cost manikin with a specific design to serve all possible needs of end users but still keep its function as necessary for training.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who hold a MD degree

Exclusion Criteria:

* Not want to complete questionnaires
* No experience in a nasal foreign body removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- In-house Manikin First, Then Market Manikin: 19 participants performed the nasal foreign body removal procedure using the in-house manikin. Later, they performed exactly the same procedure using the market manikin immediately after the in-house manikin.
- Market Manikin First, Then In-house Manikin: 18 participants performed the nasal foreign body removal procedure using the market manikin. Later, they performed exactly the same procedure using the in-house manikin immediately after the market manikin.
Period: Overall Study
Arm/Group | In-house Manikin First, Then Market Manikin | Market Manikin First, Then In-house Manikin
Started | 19 | 18
Completed | 19 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | In-house Manikin First, Then Market Manikin | Market Manikin First, Then In-house Manikin | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Median (Full Range); unit: years] | 30 [24 to 57] | 30 [24 to 57] | 30 [24 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction Scores
Description: Satisfaction scores in different manikins using a 5-point Likert scale (1-very unsatisfied to 5- very satisfied). There are a number of scale titles including proper size, proper weight, the ease of use, the ease of cleaning, the ease of maintenance, the flexibility of nasal alae relative to actual anatomy, similarity of the nasal cavity relative to actual anatomy, a well design for teaching, estimated price, participant's confidence if a manikin can upskill medical students to practice in a real patient and overall satisfaction.
Time Frame: 1 day for each manikin
Measure: Median (Full Range); unit: score on a scale
Groups:
- The In-house Manikin: participants who performed the nasal foreign body removal procedure using the in-house manikin.
- The Market Manikin: participants who performed the nasal foreign body removal procedure using the market manikin.
Arm/Group | The In-house Manikin | The Market Manikin
Number analyzed (Participants) | 37 | 37
score on a scale
  proper size | 4 [1 to 5] | 4 [1 to 5]
  proper weight | 4 [1 to 5] | 4 [1 to 5]
  the ease of use | 5 [1 to 5] | 4 [1 to 5]
  the ease of cleaning | 4 [1 to 5] | 4 [1 to 5]
  the ease of maintenance | 5 [1 to 5] | 3 [1 to 5]
  the flexibility of nasal alae | 4 [1 to 5] | 3 [1 to 5]
  similarity of nasal cavity | 4 [1 to 5] | 3 [1 to 5]
  a well design for teaching | 4 [1 to 5] | 4 [1 to 5]
  confidence that the manikin can upskill medical students | 4 [1 to 5] | 4 [1 to 5]

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- The In-house Manikin: Participants who performed nasal foreign body removal in the in-house manikin.
- The Market Manikin: Participants who performed nasal foreign body removal in market manikin.
Arm/Group | The In-house Manikin | The Market Manikin
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT04901026/Prot_SAP_000.pdf